CLINICAL TRIAL: NCT05604625
Title: A Comparison of Class Ⅱ Malocclusion Treatment Using Van Beek-headgear Activator Versus Andresen Activator: A Randomized Clinical Trial
Brief Title: Ethically Accepted With Code 851/2971 A Comparison of Class Ⅱ Malocclusion Treatment Using Van Beek-headgear Activator Versus Andresen Activator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Essam Eldein Saad Hamed Shady, doctor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 851/2971
Record Dates: First submitted 2022-10-30; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Class II Growth Modification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): 12 patients will receive Van-Beek activator and a headgear
  Interventions: Device: Van-Beek activator and a headgear
- Group B (Active Comparator): 12 patients will receive Andresen activator
  Interventions: Device: Andresen activator

INTERVENTIONS:
Device: Van-Beek activator and a headgear — 12 patients will receive Van-Beek activator and a headgear
  Arms: Group A
Device: Andresen activator — 12 patients will receive Andresen activator.
  Arms: Group B

SUMMARY:
The aim of this study is to compare the treatment results when treating Class II division 1 malocclusion using the Van Beek-Headgear Activator combination (vBHGA) appliance versus using the Andresen activator.

ELIGIBILITY:
Inclusion Criteria:

* Class II division 1 indicated by ANB angle value ≥ 4º
* Class II division 1 with overjet > 5mm.
* An age range between 8 and 13 years growing patient using cervical vertebral stage assessment (CVS).
* No previous orthodontic treatment
* No indications or symptoms of periodontal disease in the past or present, as determined by clinical and radiographic examination

Exclusion Criteria:

* Missing teeth (excluding 3rd molars).
* Craniofacial anomalies.
* Medical condition or prescription medication that may affect growth.
* Lack of compliance whenever documented in the charts.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
treating Class II division 1 malocclusion | at 8 months
  rate of mandibular and maxillary growth

CONTACTS AND LOCATIONS:
Locations (1):
- Alazhar University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Altenburger E, Ingervall B. The initial effects of the treatment of Class II, division 1 malocclusions with the van Beek activator compared with the effects of the Herren activator and an activator-headgear combination. Eur J Orthod. 1998 Aug;20(4):389-97. doi: 10.1093/ejo/20.4.389. PMID 9753820